CLINICAL TRIAL: NCT03370926
Title: (18F)-Fluoroethyl-L-tyrosine Positron Emission Tomography and Multiparametric MRI for the Delination of Target Volumes in High-grade Glioma Patients Undergoing Radiotherapy
Brief Title: FET-PET and Multiparametric MRI for High-grade Glioma Patients Undergoing Radiotherapy
Acronym: IMAGG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IMAGG
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Radiotherapy
MeSH Terms: conditions — Glioblastoma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glioblastoma is the most common malignant brain tumor in adults. The primary treatment consists of maximal tumor removal followed by radiotherapy (RT) with concomitant and adjuvant temozolomide. Tumor recurrence after chemoradiotherapy has previously been shown to be predominantly within or at the margin of the irradiated volume, but distant failure are not rare, especially in patients with MGMT methylation.Traditionally, RT has been planned based on on planning CT with co-registered postoperative MRI, with the addition of a clinical target volume margin of 2-3 cm to account for infiltrative odema.

To better characterize the disease, more specific physiological and/or metabolical markers of tumor cells, vascularization and hypoxia measured on multiparametric MRI as perfusion, diffusion and spectroscopy alongside with PET tracer like Fluoroéthyl-L-tyrosine ([18F]-FET) are now available and suggest that aggressive areas, like uptake of PET tracer and vascularity are present outside areas of contrast enhancement usually irradiated. These informations could be incorporated to optimize the treatment of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years or older
* Histologically confirmed newly diagnosed glioblastoma or anaplastic astrocytoma
* Patients must have undergone surgery with macroscopic complete resection or incomplete resection with residual disease less than 5 cm on MRI
* An MRI or a scan 48h after surgery should be available
* WHO ≤ 2
* Indication for adjuvant radiotherapy
* Surgery must have been performed 45 days before the start of radiotherapy.
* Ability to understand and to give consent

Exclusion Criteria:

* Age < 18 Years.
* Prior radiation therapy to the brain
* Any usual formal indication against MRI (claustrophobia, metallic objects or implanted medical devices in body: pacemaker, clips, prostheses ...)
* Allergic reaction to FET
* Pregnant women or nursing mothers
* Refusal to use effective contraception at study entry and throughout the study if patient is of childbearing age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with anaplastic astrocytoma or glioblastoma who are referred for adjuvant radiotherapy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Target volumes contoured on standard MRI and planning CT, FET-PET and multiparametric MRI images | 12 months
  Increase in at least 10% of irradiation target volumes compared to the result of the MRI+scanner reference technique.

SECONDARY OUTCOMES:
Treatment failure pattern in respect to the target volume based on standard MRI, multiparametric MRI and FET-PET. | 12 months
  Irradiation target volumes associated with standard MRI
Sites of failures with composite and standard MRI based RT planning | 12 months
  Irradiation target volumes associated with standard MRI based RT planning
Progression-free Survival | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Derived] Dissaux B, Mazouz Fatmi D, Ognard J, Allard B, Keromnes N, Latreche A, Lepeuve A, Schick U, Bourbonne V, Ben Salem D, Dissaux G, Querellou S. Radiotherapy Target Volume Definition in Newly Diagnosed High-Grade Glioma Using 18F-FET PET Imaging and Multiparametric MRI: An Inter Observer Agreement Study. Tomography. 2022 Aug 16;8(4):2030-2041. doi: 10.3390/tomography8040170. PMID 36006068